CLINICAL TRIAL: NCT00111007
Title: Phase III Randomized, Placebo Controlled Study of Sorafenib in Repeated Cycles of 21 Days in Combination With Paclitaxel/Carboplatin Chemotherapy in Subjects With Unresectable Stage III or Stage IV Melanoma.
Brief Title: A Treatment Combination for Patients With Unresectable Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11718; 2005-000941-12 (EudraCT Number); NCT00262912 (obsolete NCT alias)
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Sorafenib; CP protocol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Sorafenib, 400 mg orally, 2 tablets (200 mg each) bid (bis in die [twice daily]) on Study Days 2 to 19 + Paclitaxel (225 mg/m^2 iv [Intravenous]) and Carboplatin (AUC [area under the curve] 6 iv) on Study Day 1 (21 days per cycle) for double-blind (DB) treatment. Subjects who discontinued DB treatment with complete response (CR), partial response (PR) or stable disease (SD) entered active follow up period. Subjects who discontinued DB treatment with disease progression (DP) entered long term follow up period.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006); Drug: Carboplatin/Paclitaxel
- Carboplatin/Paclitaxel (C/P) (Active Comparator): Placebo, 2 tablets bid on Study Days 2-19 + Paclitaxel (225 mg/m^2 iv) and Carboplatin (AUC 6 iv) on Study Day 1 (21 days per cycle) for double-blind (DB) treatment. Subjects who discontinued DB treatment with complete response (CR), partial response (PR) or stable disease (SD) entered active follow up period. Subjects who discontinued DB treatment with disease progression (DP) entered long term follow up period.
  Interventions: Drug: Carboplatin/Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib, 400 mg po (per os), 2 tablets (200 mg each) bid Study Days 2-19
  Arms: Sorafenib (Nexavar, BAY43-9006)
Drug: Carboplatin/Paclitaxel — Paclitaxel (225 mg/m^2 iv) and Carboplatin (AUC 6 iv) on Study Day 1
Drug: Placebo — Placebo, 2 tablets bid Study Days 2-19
  Arms: Carboplatin/Paclitaxel (C/P)

SUMMARY:
The objectives of this study are to compare the anti-tumor activity as measured by Progression Free Survival (PFS) and tolerability of Sorafenib in combination with Paclitaxel and Carboplatin versus Paclitaxel and Carboplatin in combination with placebo in subjects with unresectable Stage III or Stage IV melanoma who progressed after receiving only one prior therapy containing Dacarbazine (DTIC) or Temozolomide (TMZ).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a life expectancy of at least 12 weeks
* Subjects with histologically or cytologically confirmed unresectable (Stage III) or metastatic (Stage IV) melanoma
* Subjects must have progressed after receiving at least one cycle of DTIC or TMZ containing regimen
* Subjects who have an ECOG PS of 0 or 1
* Measurable disease defined as at least one lesion that can be accurately and serially measured per the modified RECIST criteria

Exclusion Criteria:

* Primary ocular or mucosal melanoma
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta [Noninvasive papillary carcinoma], Tis [Carcinoma in situ: "flat tumor"]& T1 [Tumor invades subepithelial connective tissue]) or any cancer curatively treated < 5 years prior to study entry
* History of cardiac disease
* Known history of human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (62):
- United States (19):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Los Angeles, California
  - Aurora, Colorado
  - Tampa, Florida
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Louisville, Kentucky
  - St Louis, Missouri
  - Omaha, Nebraska
  - Montclair, New Jersey
  - Buffalo, New York
  - New York, New York
  - Columbus, Ohio
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
  - Charlottesville, Virginia
  - Seattle, Washington
- Australia (9):
  - Camperdown, New South Wales
  - Warartah, New South Wales
  - Westmead, New South Wales
  - Brisbane, Queensland
  - East Melbourne, Victoria
  - Heidelberg, Victoria
  - Malvern, Victoria
  - Melbourne, Victoria
  - Nedlands, Western Australia
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (7):
  - Bordeaux
  - Boulogne-Billancourt
  - Brest
  - Lyon
  - Montpellier
  - Paris
  - Villejuif
- Germany (10):
  - Heidelberg, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Frankfurt am Main, Hesse
  - Essen, North Rhine-Westphalia
  - Trier, Rhineland-Palatinate
  - Homburg, Saarland
  - Kiel, Schleswig-Holstein
  - Berlin, State of Berlin
- Netherlands (3):
  - Amsterdam
  - Rotterdam
  - Utrecht
- United Kingdom (9):
  - Southampton, Hampshire
  - Leicester, Leicestershire
  - London, London
  - Manchester, Manchester
  - Bebington, Merseyside
  - Nottingham, Nottinghamshire
  - Sutton, Surrey
  - Leeds, West Yorkshire
  - Swansea

REFERENCES:
- [Result] Hauschild A, Agarwala SS, Trefzer U, Hogg D, Robert C, Hersey P, Eggermont A, Grabbe S, Gonzalez R, Gille J, Peschel C, Schadendorf D, Garbe C, O'Day S, Daud A, White JM, Xia C, Patel K, Kirkwood JM, Keilholz U. Results of a phase III, randomized, placebo-controlled study of sorafenib in combination with carboplatin and paclitaxel as second-line treatment in patients with unresectable stage III or stage IV melanoma. J Clin Oncol. 2009 Jun 10;27(17):2823-30. doi: 10.1200/JCO.2007.15.7636. Epub 2009 Apr 6. PMID 19349552
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from May 4 2005 to Jan 08 2009 (first subject's first visit to last subject's last visit) at 54 centers in 7 countries: Australia (6), Canada (6), France (6), Germany (10), Netherlands (2), United Kingdom (8), and United States (16).
Pre-assignment Details: Of 315 screened subjects, 270 were randomized (45 failed screening) and were valid for Intent-To-Treat (ITT) analyses (135 in each treatment group). One subject in each group did not receive treatment: 1 died and 1 withdrew consent. Thus, 268 subjects received treatment (134 in each group) and were valid for the safety analyses.
Period: Double-blind (DB) Treatment
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Carboplatin/Paclitaxel (C/P)
Started | 135 (ITT population) | 135 (ITT population)
Received Treatment | 134 (Safety population) | 134 (Safety population)
Completed | 27 | 24
Not Completed | 108 | 111
Not completed — Adverse Event | 12 | 4
Not completed — Death | 5 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Disease progression/recurrence/relapse | 1 | 0
Not completed — Relapse | 1 | 0
Not completed — Progression by clinical judgement | 0 | 2
Not completed — Radiological and symptomatic progression | 83 | 93
Not completed — Primary reason with other category | 0 | 1
Period: Active Follow-up
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Carboplatin/Paclitaxel (C/P)
Started | 6 (Subjects discontinued DB treatment with CR, PR and SD entered this period.) | 4 (Subjects discontinued DB treatment with CR, PR and SD entered this period.)
Completed | 0 | 2
Not Completed | 6 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Death | 2 | 0
Not completed — Disease progression/recurrence/relapse | 3 | 2
Period: Long Term Follow-up
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Carboplatin/Paclitaxel (C/P)
Started | 101 (Subjects discontinued DB treatment with DP entered this period.) | 107 (Subjects discontinued DB treatment with DP entered this period.)
Completed | 54 | 62
Not Completed | 47 | 45
Not completed — Death | 34 | 39
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Disease progression/recurrence/relapse | 2 | 1
Not completed — Missing | 10 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Carboplatin/Paclitaxel (C/P) | Total
Number analyzed (Participants) | 135 | 135 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (12.8) | 55.1 (13.0) | 55.5 (57.0)
Age, Customized [Number; unit: participants]
  <65 years | 97 | 92 | 189
  65 to 74 years | 29 | 39 | 68
  >=75 years | 9 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 48 | 99
  Male | 84 | 87 | 171
American Joint Committee on Cancer (AJCC) Stage at Study Entry [Number; unit: participants] — Stage III: Clinical or radiological evidence of regional metastases (M), in either the lymph nodes or intra-lymphatic. Stage IV: M at any distant site. M1a: M to the skin, subcutaneous tissue, or lymph nodes. M1b: M to the lung. M1c: M to all other visceral sites or at any site associated with an elevated serum lactate dehydrogenase.
  participants
    Stage III or IV M1a | 16 | 11 | 27
    Stage IV M1b | 27 | 31 | 58
    Stage IV M1c | 92 | 93 | 185
Baseline Eastern Cooperative Oncology Group (ECOG) Performance [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects a patient. The scale ranges from 0 (fully active) to 5 (dead). 0=Fully active without restriction; 1= Restricted in physically strenuous activity; 2= Ambulatory, capable of all selfcare; 3= Capable of limited selfcare; 4= Completely disabled; 5= Dead. Subjects entering this study must have had an ECOG score of 0 or 1 (restricted in physically strenuous activity but ambulatory).
  participants
    Status 0 | 76 | 70 | 146
    Status 1 | 59 | 65 | 124

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was calculated as the time (days) from date of randomization to date of first observed DP (per modified Response Evaluation Criteria In Solid Tumors [RECIST] or clinical judgment, whichever was earlier: CR, PR, stable disease, progressive disease) or death due to any cause, if death occurred before progression was documented. The actual date of tumor assessments was used for this calculation. PFS for subjects without progression or death was censored at the last date of tumor evaluation. PFS for subjects who had no tumor assessments after baseline and did not die was censored at 1 day.
Time Frame: Time from randomization to documented tumor progression or death (median time of 124 days)
Population: PFS was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment. For the ITT population, subjects were included in the treatment group assigned at randomization, regardless of the treatment received.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Carboplatin/Paclitaxel (C/P)
Number analyzed (Participants) | 135 | 135
days | 122 [83 to 162] | 125 [79 to 160]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Carboplatin/Paclitaxel (C/P); Test type: Superiority or Other; p = 0.492, log rank test; Hazard Ratio (HR) = 0.906, 95% CI 2-sided [0.627 to 1.310]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was calculated as the number of days from date of randomization to death date. Subjects who had not died at the time of analysis were censored at their last contact date.
Time Frame: Time from randomization to death (median time of 294 days)
Population: OS was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment. For the ITT population, subjects were included in the treatment group assigned at randomization, regardless of the treatment received.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Carboplatin/Paclitaxel (C/P)
Number analyzed (Participants) | 135 | 135
days | 294 [247 to 321] | 294 [259 to 382]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Carboplatin/Paclitaxel (C/P); Test type: Superiority or Other; p = 0.979, log rank test; Hazard Ratio (HR) = 0.996, 95% CI 2-sided [0.744 to 1.333]

3. Secondary Outcome: Time to Progression (TTP)
Description: TTP was calculated as the time (days) from date of randomization to date of first observed disease progression (DP) (per modified RECIST or clinical judgment, whichever was earlier: CR, PR, stable disease, progressive disease). The actual dates of tumor assessments were used for this calculation. TTP for subjects without disease progression at the time of analysis, including subjects with death prior to progression, was censored at the last date of tumor evaluation. TTP for subjects who had no tumor assessments after baseline was censored at 1 day.
Time Frame: Time from randomization to documented tumor progression (median time of 126 days)
Population: TTP was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment. For the ITT population, subjects were included in the treatment group assigned at randomization, regardless of the treatment received.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Carboplatin/Paclitaxel (C/P)
Number analyzed (Participants) | 135 | 135
days | 126 [90 to 167] | 126 [83 to 160]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Carboplatin/Paclitaxel (C/P); Test type: Superiority or Other; p = 0.331, log rank test; Hazard Ratio (HR) = 0.863, 95% CI 2-sided [0.641 to 1.162]

4. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined as the time from the first documented objective response of Partial Response (PR: At least a 30% decrease in the sum of the longest diameter [SLD] of target lesions, taking as reference the baseline SLD or better) or Complete Response (CR: Disappearance of all target lesions), whichever was noted earlier, to disease progression or death (if death occurred before progression was documented). Duration of response for subjects who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment.
Time Frame: Time from initial response to documented tumor progression or death (median time of 197 days)
Population: DOR was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment. For the ITT population, subjects were included in the treatment group assigned at randomization, regardless of the treatment received.
Measure: Median (Full Range); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Carboplatin/Paclitaxel (C/P)
Number analyzed (Participants) | 135 | 135
days | 228 [42 to 420] | 166 [46 to 209]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Carboplatin/Paclitaxel (C/P); Test type: Superiority or Other; p = 0.146, log rank test; Hazard Ratio (HR) = 0.398, 95% CI 2-sided [0.110 to 1.437]

5. Secondary Outcome: Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status to the Visit When the Best Tumor Response Was Noted
Description: Change in ECOG PS is defined as an improvement (increase) or worsening (decrease) of at least one grade from the baseline ECOG score (from 0 [fully active] to 5 [dead]). Change in ECOG PS was recorded at the visit at which best confirmed response (BCR) using the modified RECIST (PR, CR, stable disease or Progressive Disease (PD)) was first noted (the change was 7% for both Sorafenib and Placebo). The BCR is the BCR recorded from the start of the treatment until DP/recurrence (taking as reference for DP, the smallest measurements recorded since treatment started).
Time Frame: baseline and at visit when best response was noted (maximum treatment duration of 68.3 weeks)
Population: Change in ECOG PS was analyzed for the intent to treat (ITT) population, defined as all subjects randomized to treatment. For the ITT population, subjects were included in the treatment group assigned at randomization, regardless of the treatment received.
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Carboplatin/Paclitaxel (C/P)
Number analyzed (Participants) | 135 | 135
participants
  missing | 10 | 4
  better | 9 | 10
  no change | 70 | 82
  worse | 46 | 39
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Carboplatin/Paclitaxel (C/P); Test type: Superiority or Other; p = 0.389, Fisher Exact

ADVERSE EVENTS:
Description: Abbreviations used in the Adverse Events section: Absolute Neutrophil Count (ANC), Aspartate Aminotransferase (AST), Central Nervous System (CNS), Common Terminology Criteria for Adverse Events (CTCAE), Gastro-Intestinal (GI), Genito-Urinary (GU), National Cancer Institute (NCI), Not Otherwise Specified (NOS)
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Carboplatin/Paclitaxel (C/P)
Serious Adverse Events (participants affected / at risk) | 66/134 | 65/134
Other Adverse Events (participants affected / at risk) | 132/134 | 134/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=134) | Carboplatin/Paclitaxel (C/P) (N=134)
allergic reaction (Immune system disorders) | 4 | 2
neutrophils (Blood and lymphatic system disorders) | 15 | 7
hemoglobin (Blood and lymphatic system disorders) | 3 | 8
platelets (Blood and lymphatic system disorders) | 0 | 3
leukocytes (Blood and lymphatic system disorders) | 2 | 1
supraventricular arrhythmia, atrial flutter (Cardiac disorders) | 1 | 1
supraventricular arrhythmia, supraventricular extrasystoles (pac; premature nodal/junction contr) (Cardiac disorders) | 0 | 1
supraventricular arrhythmia, supraventricular arrhythmia NOS (Cardiac disorders) | 1 | 0
tachycardia (Cardiac disorders) | 0 | 1
vasovagal episode (Cardiac disorders) | 0 | 1
hypotension (Cardiac disorders) | 1 | 2
cardiac ischemia / infarction (Cardiac disorders) | 2 | 0
cardiac general - other (Cardiac disorders) | 0 | 0
left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1
pericarditis (Cardiac disorders) | 0 | 1
death not associated with CTCAE term, disease progression NOS (General disorders) | 2 | 1
death not associated with CTCAE term, death NOS (General disorders) | 1 | 0
diabetes (Endocrine disorders) | 1 | 0
fever (General disorders) | 3 | 5
fatigue (General disorders) | 2 | 4
constitutional symptoms - other (General disorders) | 1 | 4
vomiting (Gastrointestinal disorders) | 1 | 4
diarrhea (Gastrointestinal disorders) | 2 | 2
dehydration (Gastrointestinal disorders) | 1 | 2
obstruction, GI, small bowel NOS (Gastrointestinal disorders) | 1 | 2
anorexia (Gastrointestinal disorders) | 0 | 2
constipation (Gastrointestinal disorders) | 2 | 0
nausea (Gastrointestinal disorders) | 1 | 1
colitis (Gastrointestinal disorders) | 0 | 1
esophagitis (Gastrointestinal disorders) | 0 | 1
fistula, GI, esophagus (Gastrointestinal disorders) | 0 | 1
CNS hemorrhage (Vascular disorders) | 2 | 2
hemorrhage - other (Vascular disorders) | 1 | 1
hemorrhage, GI, lower GI NOS (Vascular disorders) | 0 | 1
hemorrhage with surgery (Vascular disorders) | 1 | 0
hemorrhage pulmonary, respiratory tract NOS (Vascular disorders) | 1 | 0
hemorrhage, GU, bladder (Vascular disorders) | 0 | 1
hemorrhage, GU, urinary NOS (Vascular disorders) | 0 | 1
liver dysfunction (Hepatobiliary disorders) | 1 | 1
cholecystitis (Hepatobiliary disorders) | 1 | 0
febrile neutropenia (Infections and infestations) | 10 | 8
infection with unknown ANC, lung (pneumonia) (Infections and infestations) | 1 | 3
infection with unknown ANC, skin (cellulitis) (Infections and infestations) | 2 | 1
infection with normal ANC, upper airway NOS (Infections and infestations) | 1 | 1
infection - other (Infections and infestations) | 0 | 2
infection (documented clinically), upper airway NOS (Infections and infestations) | 1 | 0
infection with normal ANC, blood (Infections and infestations) | 0 | 1
infection with normal ANC, lung (pneumonia) (Infections and infestations) | 0 | 1
infection with normal ANC, soft tissue NOS (Infections and infestations) | 0 | 1
infection with normal ANC, vein (Infections and infestations) | 1 | 0
infection with normal ANC, wound (Infections and infestations) | 0 | 1
muscle weakness, whole body / generalized (Musculoskeletal and connective tissue disorders) | 1 | 0
hyperglycemia (Metabolism and nutrition disorders) | 0 | 3
AST (Metabolism and nutrition disorders) | 0 | 1
hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
hyponatremia (Metabolism and nutrition disorders) | 1 | 0
seizure (Nervous system disorders) | 1 | 6
confusion (Nervous system disorders) | 0 | 2
neuropathy: motor (Nervous system disorders) | 2 | 0
CNS ischemia (Nervous system disorders) | 1 | 0
speech impairment (Nervous system disorders) | 1 | 0
neurology - other (Nervous system disorders) | 0 | 1
neuropathy: sensory (Nervous system disorders) | 1 | 0
somnolence (Nervous system disorders) | 1 | 0
syncope (fainting) (Nervous system disorders) | 0 | 1
pain, abdomen NOS (General disorders) | 2 | 4
pain, pain NOS (General disorders) | 3 | 1
pain, chest / thorax NOS (General disorders) | 2 | 0
pain, tumor pain (General disorders) | 0 | 1
pain, joint (General disorders) | 1 | 0
pain, muscle (General disorders) | 0 | 1
dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 2
pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 1 | 1
aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
hand - foot skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
rash / desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
thrombosis / thrombus / embolism (Vascular disorders) | 3 | 9
no code in CTCAE (General disorders) | 1 | 0
intraop injury, bone (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=134) | Carboplatin/Paclitaxel (C/P) (N=134)
allergic reaction (Immune system disorders) | 8 | 10
neutrophils (Blood and lymphatic system disorders) | 68 | 71
platelets (Blood and lymphatic system disorders) | 62 | 40
hemoglobin (Blood and lymphatic system disorders) | 33 | 44
leukocytes (Blood and lymphatic system disorders) | 36 | 38
lymphopenia (Blood and lymphatic system disorders) | 8 | 5
hypertension (Cardiac disorders) | 11 | 6
fatigue (General disorders) | 102 | 79
insomnia (General disorders) | 26 | 25
fever (General disorders) | 16 | 11
sweating (General disorders) | 10 | 16
weight loss (General disorders) | 16 | 9
rigors / chills (General disorders) | 10 | 8
constitutional symptoms - other (General disorders) | 3 | 7
nausea (Gastrointestinal disorders) | 71 | 72
diarrhea (Gastrointestinal disorders) | 64 | 36
constipation (Gastrointestinal disorders) | 40 | 42
vomiting (Gastrointestinal disorders) | 33 | 32
anorexia (Gastrointestinal disorders) | 32 | 15
mucositis (functional / symptomatic), oral cavity (Gastrointestinal disorders) | 17 | 11
taste alteration (Gastrointestinal disorders) | 11 | 13
heartburn (Gastrointestinal disorders) | 12 | 11
GI - other (Gastrointestinal disorders) | 13 | 6
dry mouth (Gastrointestinal disorders) | 7 | 3
flatulence (Gastrointestinal disorders) | 7 | 3
hemorrhage pulmonary, nose (Vascular disorders) | 18 | 10
infection - other (Infections and infestations) | 7 | 8
infection with normal ANC, upper airway NOS (Infections and infestations) | 7 | 6
infection with unknown ANC, skin (cellulitis) (Infections and infestations) | 7 | 0
edema: limb (Blood and lymphatic system disorders) | 14 | 18
musculoskeletal - other (Musculoskeletal and connective tissue disorders) | 8 | 6
hypokalemia (Metabolism and nutrition disorders) | 9 | 11
hypomagnesemia (Metabolism and nutrition disorders) | 5 | 10
hypophosphatemia (Metabolism and nutrition disorders) | 8 | 4
lipase (Metabolism and nutrition disorders) | 7 | 3
neuropathy: sensory (Nervous system disorders) | 89 | 87
dizziness (Nervous system disorders) | 21 | 19
mood alteration, depression (Nervous system disorders) | 9 | 11
neuropathy: motor (Nervous system disorders) | 7 | 5
neurology - other (Nervous system disorders) | 8 | 4
blurred vision (Eye disorders) | 8 | 11
pain, joint (General disorders) | 44 | 37
pain, muscle (General disorders) | 35 | 27
pain, extremity - limb (General disorders) | 25 | 23
pain, abdomen NOS (General disorders) | 19 | 23
pain, head / headache (General disorders) | 21 | 20
pain, back (General disorders) | 12 | 18
pain, bone (General disorders) | 13 | 17
pain, pain NOS (General disorders) | 13 | 12
pain, throat / pharynx / larynx (General disorders) | 11 | 6
pain, chest / thorax NOS (General disorders) | 10 | 5
cough (Respiratory, thoracic and mediastinal disorders) | 29 | 25
dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 20 | 24
voice changes (Respiratory, thoracic and mediastinal disorders) | 10 | 4
hiccoughs (Respiratory, thoracic and mediastinal disorders) | 9 | 4
pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 4 | 9
alopecia (Skin and subcutaneous tissue disorders) | 90 | 87
rash / desquamation (Skin and subcutaneous tissue disorders) | 79 | 29
hand - foot skin reaction (Skin and subcutaneous tissue disorders) | 38 | 8
pruritus (Skin and subcutaneous tissue disorders) | 34 | 12
dermatology - other (Skin and subcutaneous tissue disorders) | 19 | 6
dry skin (Skin and subcutaneous tissue disorders) | 16 | 5
erythema multiforme (Skin and subcutaneous tissue disorders) | 12 | 8
flushing (Skin and subcutaneous tissue disorders) | 6 | 7
injection site reaction (Skin and subcutaneous tissue disorders) | 7 | 5
acne (Skin and subcutaneous tissue disorders) | 1 | 9
urticaria (Skin and subcutaneous tissue disorders) | 8 | 1

LIMITATIONS AND CAVEATS:
Metastatic melanoma is notorious for its resistance to chemotherapy. Thus, it is unlikely that inhibition of a single factor or pathway would produce a sustained clinical effect in patients with previously treated, highly refractory disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less